CLINICAL TRIAL: NCT07344597
Title: Prospective Comparative Study of Hypofractionated Adjuvant Radiotherapy in 2 Virsus 3 Weeks in Breast Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Salwa Shawky Bakeet Ali (Other)
Responsible Party: Sponsor-Investigator, Salwa Shawky Bakeet Ali, assiut, Assiut University
Organization: Assiut University (Other)
Other Study IDs: adjuvant radiotherapy in BC
Record Dates: First submitted 2025-09-25; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A: hypofractionated adjuvant radiotherapy regimens 40.05 Gy in 15 fractions in breast cancer in 3w
  Interventions: Device: radiotherapy
- B: hypofractionated adjuvant radiotherapy regimens 34 Gy in 10
  fractions in 2w
  Interventions: Device: radiotherapy

INTERVENTIONS:
Device: radiotherapy — Hypofractionated Adjuvant Radiotherapy in 2 versus 3 Weeks of Breast Cancer and effect skin toxicity and over all survival

SUMMARY:
To compare the efficacy and safety of two hypofractionated adjuvant radiotherapy regimens 34 Gy in 10

fractions versus 40.05 Gy in 15 fractions in patients with breast cancer treated at the South Egypt Cancer

Institute.

DETAILED DESCRIPTION:
Female breast cancer (BC) has been the leading cause of cancer morbidity and mortality among women in the

majority of countries for decades. In 2020, there were an estimated 2.3 million new cases and 685,000 deaths

from female BC worldwide, which accounted for one in four cancer cases and one in six cancer deaths among

women.

u For women with newly diagnosed, non-metastatic breast cancer, treatment consists of a multidisciplinary

approach that involves input from surgery, radiation oncology, and medical oncology. The objective of adjuvant

radiation therapy (RT) is to eradicate any tumor deposits remaining following surgery for patients treated by

either breast-conserving surgery or mastectomy . Doing so reduces risk of locoregional recurrence and improves

breast cancer-specific and overall survivals.

u A historical regimen of 25-28 fractions over 6 weeks was adopted for radiotherapy (RT) following breast-

conserving surgery (BCS) and total mastectomy. An early assumption that breast cancer cell lines might be more

sensitive to fractional doses than acute skin reactions and other squamous carcinomas lead to development of the

hypofractionated RT (HypoRT) approach, which elevated fractional dose up to 3 Gy with reduced total

dose/fractions, for obtaining radiobiological equivalence to a traditional regimen of 50-50.4 Gy in 25-28

fractions.

u Recently, the American Society of Radiation Oncology released a task force guideline recommending

hypofractionated radiotherapy for all women of any age whether they had received chemotherapy or not ,Their

evidence-based recommendations were supported by studies from Canada and the United Kingdom.

u Benefits of HypoRT include both, radiobiologic advantages and reduced length of treatment courses, for

improving healthcare resources and patient convenience. Consequently, HypoRT has been widely adopted

worldwide based on a series of randomized clinical trials .

u Recently, HypoRT over 3 weeks and with shorter courses of 5 fractions have been recommended in treatment

guidelines.

u Regarding clinical outcomes of a 2-week fractionation schedule , it was observed that acute and late effects were

acceptable with control rates similar to those reported in other trials with hypofractionation,Based

on these findings we started a trial to compare a 3-week radiotherapy schedule with a 2-week schedule .

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥18 years.

Female or male patients with invasive carcinoma of the breast.

Complete microscopic excision of primary tumor.

Undergoing breast-conserving surgery (BCS) or modified radical mastectomy (MRM).

≥ Axillary lymph nodes dissected.

T1_4pN0_3M0 disease.

Neoadjuvant or adjuvant CTH .

Signed informed consent and able to comply with follow up.

Exclusion Criteria:

* Evidence of distant metastases.

Past history of malignancy.

Prior radiotherapy to the chest region

Simultaneous malignancy (except non-melanoma skin cancer or in situ cervical carcinoma)

Connective tissue diseases (e.g., lupus erythematosus, scleroderma)

Pregnancy or lactation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: breast cancer patients above 18y,with invasive carcinoma,excision of primary,recieved neoadjuvant or adj cth .
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Disease free survival analyzed from the date of diagnosis. | through study completion, an average of 1 year
  local control was defined as absence of disease in the irradiated areas.recurrence were categorized as local(breast or surgical bed), regional(lymphatic drainage of axillary, supraclavicular fossa or internal mammary chain),or distant (metastasis),and any associayion of these

SECONDARY OUTCOMES:
Assessment of Acute Skin Toxicity | From start of radiotherapy through 3 months after completion of radiotherapy
  Acute toxicities will be assessed according to RTOG criteria. The most severe toxicity presented will be reported.
Assessment of Late Skin Toxicity | From 3 months after completion of radiotherapy through study completion, an average of 1 year
  Late toxicities will be assessed according to RTOG criteria. The most severe toxicity presented will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit, Asyut, Egypt

REFERENCES:
- [Result] Youssef A, Stanford J. Hypofractionation Radiotherapy vs. Conventional Fractionation for Breast Cancer: A Comparative Review of Toxicity. Cureus. 2018 Oct 29;10(10):e3516. doi: 10.7759/cureus.3516. PMID 30648051
- [Result] Eraso A, Sanz J, Molla M, Reyes V, Pedro A, Arenas M, Martinez E, Ballester R, Cambra MJ, Garcia V, Prades JL, Borras JM, Algara M. Evidence-based guidelines for hypofractionated radiation in breast cancer: conclusions of the Catalan expert working group. Clin Transl Oncol. 2022 Aug;24(8):1580-1587. doi: 10.1007/s12094-022-02798-8. Epub 2022 Feb 21. PMID 35190961
- [Result] Kim N, Kim YB. Journey to hypofractionation in radiotherapy for breast cancer: critical reviews for recent updates. Radiat Oncol J. 2022 Dec;40(4):216-224. doi: 10.3857/roj.2022.00577. Epub 2022 Dec 26. PMID 36606299
- [Result] Yadav BS, Dahiya D, Gupta A, Rana D, Robert N, Sharma M, Rao B. Breast cancer hypofractionated radiotherapy in 2-weeks with 2D technique: 5-year clinical outcomes of a phase 2 trial. Rep Pract Oncol Radiother. 2021 Aug 12;26(4):503-511. doi: 10.5603/RPOR.a2021.0054. eCollection 2021. PMID 34434565
- [Result] START Trialists' Group; Bentzen SM, Agrawal RK, Aird EG, Barrett JM, Barrett-Lee PJ, Bliss JM, Brown J, Dewar JA, Dobbs HJ, Haviland JS, Hoskin PJ, Hopwood P, Lawton PA, Magee BJ, Mills J, Morgan DA, Owen JR, Simmons S, Sumo G, Sydenham MA, Venables K, Yarnold JR. The UK Standardisation of Breast Radiotherapy (START) Trial A of radiotherapy hypofractionation for treatment of early breast cancer: a randomised trial. Lancet Oncol. 2008 Apr;9(4):331-41. doi: 10.1016/S1470-2045(08)70077-9. Epub 2008 Mar 19. PMID 18356109
- [Result] Zhang Y, Ji Y, Liu S, Li J, Wu J, Jin Q, Liu X, Duan H, Feng Z, Liu Y, Zhang Y, Lyu Z, Song F, Song F, Yang L, Liu H, Huang Y. Global burden of female breast cancer: new estimates in 2022, temporal trend and future projections up to 2050 based on the latest release from GLOBOCAN. J Natl Cancer Cent. 2025 Feb 13;5(3):287-296. doi: 10.1016/j.jncc.2025.02.002. eCollection 2025 Jun. PMID 40693239